CLINICAL TRIAL: NCT05489952
Title: Efficacy and Safety of Perioperative Iron Supplementation for Postoperative Rehabilitation of Geriatric Hip Fractures: a Multicenter, Randomized, Controlled Trial.
Brief Title: Iron Supplementation for Geriatric Hip Fractures
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: He Qifei (Other)
Responsible Party: Sponsor-Investigator, He Qifei, Principal Investigator, Shenzhen Second People's Hospital
Organization: Shenzhen Second People's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20223357010
Record Dates: First submitted 2022-07-31; First posted 2022-08-05 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Hip Fractures; Fragility Fracture; Osteoporotic Fractures
MeSH Terms: conditions — Hip Fractures; Osteoporotic Fractures | interventions — Ferric Oxide, Saccharated; ferrous lactate

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- iron supplement group (Experimental)
  Interventions: Drug: iron sucrose and ferrous lactate
- control group (No Intervention)

INTERVENTIONS:
Drug: iron sucrose and ferrous lactate — The experimental group added to the intravenous iron sucrose during perioperative period according to the degree of iron deficiency. If there is still a iron deficiency or anemia at discharge, oral ferrous lactate is added after discharge.
  Other Names: iron supplementation
  Arms: iron supplement group

SUMMARY:
Geriatric hip fracture is an important disease that affects the health life of the elderly in China. Geriatric hip fracture is often complicated by a variety of comorbidities due to advanced age. And anemia is a common comorbidity. At present perioperative management of geriatric hip fracture, transfusion is only indicated for moderate and severe anemia, while no special medical intervention for mild anemia in China. More and more studies have found that iron can not only correct anemia, but also improve cardiac function, patients' quality of life and function. This study investigated the effect of perioperative iron supplementation on activity tolerance in elderly patients with hip fracture complicated with iron deficiency anemia. The study was a randomized, parallel controlled clinical study. Due to the requirements of the ethics committee, the unblinded setting was cancelled due to ethical considerations. Research will be grouped according to whether to accept iron supplementation treatment, are divided into 2 groups, respectively, iron treatment group and the traditional method. The method of randomization was stratified block randomization. The experimental group added to the intravenous iron sucrose during perioperative period according to the degree of iron deficiency. If there is still a iron deficiency or anemia at discharge, oral ferrous lactate is added after discharge. The outcomes include 6-minute walk distance, Harris score, EQ-5D score six months after surgery, perioperative blood transfusion rate, and so on in the two groups.

ELIGIBILITY:
Inclusion Criteria:

1. >65 years old patients with hip fracture
2. Patients with iron deficiency or anemia,

   * preoperative hemoglobin <13g/ dL in males and <12g/ dL in females, and >9g/ dL,
   * serum ferritin < 100 ng/ mL or serum ferritin 100-299 ng/ mL or transferrin saturation (TSAT) <20%

Exclusion Criteria:

1. Coronary artery bypass grafting, percutaneous transluminal coronary angioplasty, and cardiac device implantation (including cardiac resynchronization) within preoperative 30 days
2. Acute coronary syndrome, transient ischemic attack or stroke occurred within 30 days before surgery;
3. Refused to sign the consent form to be included in the clinical trial group;
4. Can't walk before injury;
5. Use erythropoietic preparation within 3 months before surgery and oral iron preparation within 4 weeks 30 days before surgery(> 100 mg/ day)
6. Patients with liver and kidney dysfunction
7. Other conditions that the researchers considered inappropriate for inclusion

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 444 (Estimated)
Dates: Start 2022-09-15 (Estimated); Primary Completion 2025-02-15 (Estimated); Study Completion 2025-08-15 (Estimated)

PRIMARY OUTCOMES:
6-minute walk distance | 6 months
  The 6-minute walk distance (6 MWD) provides a measure for integrated global response of multiple cardiopulmonary and musculoskeletal systems involved in exercise. The 6 MWT provides information regarding functional capacity, response to therapy and prognosis across a broad range of chronic cardiopulmonary conditions.

SECONDARY OUTCOMES:
Harris hip score | 6 months
  The Harris Hip Scale (HHS) was developed for the assessment of the results of hip surgery, and is intended to evaluate various hip disabilities and methods of treatment in an adult population.
perioperative blood transfusion rate | 1 week
  The proportion of the transfusions number to the total number of patients

CONTACTS AND LOCATIONS:
Locations (1):
- Shenzhen Second People's Hospita, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided